CLINICAL TRIAL: NCT03769389
Title: Assessing the Glycaemic Index of Two Different Cultivars of Date Fruit When Mixed With 0% Fat Yogurt on Healthy Volunteers.
Brief Title: Assessing the Glycaemic Index of Two Different Cultivars of Date Fruit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DFGI
Record Dates: First submitted 2018-03-27; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: GI Glycaemic Index Healthy Volunteers; GL Glycaemic Load Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- assessing the GI + GL of Birhi + YEO 0% fat yoghurt (Experimental): 47g of total carbohydrate in which contains 43.6g of Freeze-dried of Birhi powder+ 150g of 0% fat yoghurt
  Interventions: Dietary Supplement: Birhi; Dietary Supplement: Khassab; Dietary Supplement: placebo
- assessing the GI + GL of Khassab + YEO 0% fat yoghurt (Experimental): 47g of total carbohydrate in which contains34.6g of freeze-dried Khassab powder+ 150g of 0% fat yoghurt
  Interventions: Dietary Supplement: Birhi; Dietary Supplement: Khassab; Dietary Supplement: placebo
- assessing the GI + GL of 50g of Glucose in 100 ml of water (Experimental): 50g of pure glucose dissolved in 100ml of water
  Interventions: Dietary Supplement: Birhi; Dietary Supplement: Khassab; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Birhi — Birhi which contain the following:
  43.6g of Freeze-dried date powder+ 150g of 0% fat yoghurt
Dietary Supplement: Khassab — 34.6g of freeze-dried date powder+ 150g of 0% fat yoghurt
Dietary Supplement: placebo — 50g of pure glucose dissolved in 100ml of water

SUMMARY:
Fruit of the date palm (P. dactylifera) may be considered as an emerging and potential candidate for the development of health-promoting foods, owing to its high nutritional values.

Furthermore, aqueous extracts of dates have previously been shown to have potent antioxidant activity, because they inhibit in vitro lipid and protein oxidation and possess free radical scavenging capacity.

Although the high sugar content of date fruit has always been a concern, date fruit has been regarded as a low-GI to medium-GI food. However, very limited, inconsistent and contradictory information is available on the glycaemic index values of different date varieties, which may be attributed to both the methodology as well as other food factors. Date consumption is high among people of Arabic origin, where it's very common for them to be eaten with coffee or yoghurt. Therefore, in view of these concerns, the objective of this trial is to evaluate the glycaemic response of two different varieties of dates, named Birhi & Khassab, in an early maturation stage (Rutab stage), when mixed with 0% fat yogurt, on ten healthy participants aged between 18 and 45.

DETAILED DESCRIPTION:
Introduction Although, the fruit of the date palm (P. dactylifera) may be considered an emerging and potential candidate for the development of health-promoting foods owing to its high nutritive values,the high sugar content of date fruit has always been a concern. Sun-dried dates, which is the well-known ripening stage of date fruit, can be regarded as low-GI to medium-GI food. However, very limited, inconsistent and contradictory information is available on the glycaemic Index values of different date varieties. This variation could be attributed to either the methodology or the food factors.

Rational and objective Nowadays, low-GI foods have often been found to induce beneficial effects on risk factors for certain non-communicable chronic diseases . As the chemical composition of dates can vary depending on cultivar, soil conditions, agronomic practices as well as the ripening stage. It is important to know the GI of the local/regional date varieties, and in different date products such as dates with yoghurt. Date consumption is high among people of Arabic origin, where it is very commonly eaten with coffee or yoghurt. During the first trial of this PHD project, treatments containing 150g of 0% fat yoghurt and two different freeze dried date powders, depending on if it was a Birhi treatment or Khassab treatment, were formulated. These were used to assess acute effects of date fruit and yoghurt on mood and cognitive performance in healthy volunteers, as per the ethical approval from Newcastle University. These exact treatments will be used again, and the trial will aim to evaluate their glycaemic index on 10 healthy participants.

Participants Ten healthy participants aged between 18 and 45 will be recruited. Participants will be required to undergo a screening visit, followed by three study visits, which will last 2:15 minutes for each visit. Glycaemic indexes will be calculated using standard methods. Results will be calculated using means and standard deviations.

Design

A standard experimental study involving the measurement of the glycaemic responses of the ingestion of two different varieties of dates, when mixed with 0% fat yoghurt, and a placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants A total of 10 healthy participants aged between 18 and 45 will be recruited through advertisement via poster and flyer. This is an internationally recognised standard protocol which recommends using 10 volunteers or replicates for each foodstuff, and all participants will be required to undergo a screening visit.

Inclusion Criteria Healthy participants aged 18-45 with a BMI >18 <36 will be recruited from the Newcastle Upon-Tyne area.

Exclusion Criteria:

Participants will be considered ineligible to participate in the study if they meet any of the following criteria:

1. They have any metabolic diseases such as type 1 or type 2 diabetes.
2. They have a BMI above 35kg/m2 or lower than 18kg/m2
3. They are taking any illicit or prescribed drugs.
4. They are using dietary supplements, over the counter medicine or recreational drugs
5. They are females who are pregnant or seeking to become pregnant.
6. They have allergies to any food products.
7. They have any dairy intolerances.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentrations (mml/15 min)after the consumption Birhi | Change from baseline BG level at minute 15,30,45,60,75,90,105, 120 post dose
  On each of the study days, blood glucose will be measured at baseline, 15 min post-dose, 30 min post-dose, 45 min post-dose, 60 min post-dose, 75 min post-dose, 90 min post-dose, 105 min post-dose and 120 min post- dose.
Blood glucose concentrations (mml/15 min)after the consumption Khassab | Change from baseline BG level at minute 15,30,45,60,75,90,105, 120 post dose
  On each of the study days, blood glucose will be measured at baseline, 15 min post-dose, 30 min post-dose, 45 min post-dose, 60 min post-dose, 75 min post-dose, 90 min post-dose, 105 min post-dose and 120 min post- dose.
Blood glucose concentrations (mml/15 min)after the consumption Placebo | Change from baseline BG level at minute 15,30,45,60,75,90,105, 120 post dose
  On each of the study days, blood glucose will be measured at baseline, 15 min post-dose, 30 min post-dose, 45 min post-dose, 60 min post-dose, 75 min post-dose, 90 min post-dose, 105 min post-dose and 120 min post- dose.

CONTACTS AND LOCATIONS:
Locations (1):
- NU-Food Research Facility, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided